CLINICAL TRIAL: NCT02252874
Title: Can Entertaining Action-video Games Enhance Dynamic Visual Functions and Improve Balance? A Randomized Controlled Trial.
Brief Title: Can Entertaining Action-video Games Enhance Dynamic Visual Function and Improve Balance? A Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: University of Waterloo (Other); University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Allen MY Cheong, Phd, Assistant Professor, School of Optometry, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: K-ZK 93
Record Dates: First submitted 2014-09-24; First posted 2014-09-30 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Vision, Balance and Falls in Older Adults
Keywords: balance; visual function; community-dwelling older adults; action video-game

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Placebo Comparator): Receive leisure activities (e.g. reading, web-surfing, playing chess/ Mahjong) Twenty hours (2-3 sessions per week, 1.5 hours per session)
  Interventions: Behavioral: Control
- Intervention Group 1 (Active Comparator): Receive slow motion Nintendo Wii video games Twenty hours ( 2-3 sessions per week, 1.5 hours per session)
  Interventions: Behavioral: Slow-paced action video game
- Intervention Group 2 (Active Comparator): Receive fast motion Nintendo Wii video games (e.g. shooting game) Twenty hours ( 2-3 sessions per week, 1.5 hours per session)
  Interventions: Behavioral: Fast-paced action video game

INTERVENTIONS:
Behavioral: Slow-paced action video game — 20 hours slow-paced action video games
  Arms: Intervention Group 1
Behavioral: Fast-paced action video game — 20 hours fast-paced action video games
  Arms: Intervention Group 2
Behavioral: Control — 20 hours leisure activities
  Arms: Control Group

SUMMARY:
This project is aimed to find out whether action video games can enhance dynamic visual function and improve balance function in the community-dwelling older adults. It is also aimed to examine the relationship between dynamic visions and balance functions.

DETAILED DESCRIPTION:
Balance control is an important component even in a very simple daily task like walking. However, as we age, our physical and visual function would gradually deteriorate even in the absence of health or eye problems. Improving elderly balance control through different training is one way to prevent falls. In our project, we investigate the use of action video games, which is easy-to-find and entertaining, as a visual function trainer to improve balance of older adults.

We hypothesize that the training would show an improvement in both balance and dynamic vision. Our primary hypothesis is that postural sway in static and dynamic balance measures will improve after action video-game intervention. For secondary outcome measures, we hypothesize that the training will improve dynamic visual function (as measured by dynamic visual acuity and dynamic contrast sensitivity), and visual attention measures (as measured by useful field of view, multiple object tracking and spatial attention).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and speak Cantonese
* No formal training or regular practice of balance function (e.g. Tai-chi)
* Little and preferably no video-game experience
* Best corrected distance acuity of 0.2 logMAR or better

Exclusion Criteria:

* Any diagnosed ocular diseases and ocular-motor abnormalities
* Suffering form severe medical problems or self reported neurological or cognitive disorders
* Suffering from physical impairments or physical limitations restricting them from training
* Having self reported vestibular or cerebellar dysfunction, history of vertigo or severe hearing loss
* Suffering from crippling arthritis, or a recent fracture of lower limb
* Planned major surgery during the trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-09; Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Static and dynamic postural sway on forced platform | Change from baseline at week 8 and change from baseline at week 16
  1. Static Balance - postural sway when standing on firm or foam surface.
  2. Dynamic Balance:
     1. Limits of stability (LOS)
     2. Sequential weight shifting test (SWS)

SECONDARY OUTCOMES:
Grating visual acuity at different moving speeds | Change from baseline at week 8 and change from baseline at week 16
  Dynamic visual function measure - Grating visual acuity is measured with different moving speeds
Useful Field of View (UFOV) | Change from baseline at week 8 and change from baseline at week 16
  One of the visual attention measures - Useful Field of View (UFOV)
Multiple tracking objects (MOT) | Change from baseline at week 8 and change from baseline at week 16
  One of the visual attention measures - Multiple tracking objects (MOT)

CONTACTS AND LOCATIONS:
Overall Officials: Allen MY Cheong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Allen MY Cheong, Hong Kong, China